CLINICAL TRIAL: NCT00665834
Title: Comparison of the Effect Noted in The Apo/Apo-1 Ratio Using Rosuvastatin and Atorvastatin in Patients With acUte Coronary Syndrome CENTAURUS Study
Brief Title: Comparison of Rosuvastatin and Atorvastatin in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Stephen LaHaye, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMED 938-06
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Dyslipidemia; Acute Coronary Syndromes
MeSH Terms: conditions — Dyslipidemias; Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Rosuvastatin 20 mg versus placebo 20 mg
  Interventions: Drug: rosuvastatin; Drug: placebo
- 2 (Active Comparator): rosuvastatin 20 mg versus atorvastatin 80 mg
  Interventions: Drug: rosuvastatin; Drug: atorvastatin

INTERVENTIONS:
Drug: rosuvastatin — rosuvastatin 20 mg from day 0 to (maximum) day 6
  Arms: 1
Drug: placebo — placebo 20 mg from day 0 to (maximum) day 6
  Arms: 1
Drug: rosuvastatin — rosuvastatin 20 mg from discharge until the end of the study
  Arms: 2
Drug: atorvastatin — atorvastatin 80 mg from discharge until the end of the study
  Arms: 2

SUMMARY:
This is a 3-month, randomized, parallel-group study with 2 periods, comparing the efficacy and the safety of rosuvastatin 20 mg versus atorvastatin 80 mg in patients with an acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
Patients with ACS (acute coronary syndrome) constitute a high-risk population with unstable coronary disease (CHD) that differs from stable CHD primarily in short term prognosis (prediction of outcome). The 1-year rate of death or non-fatal MI (myocardial infarction or heart attack) was 13% in patients with ACS in a recent controlled study (FRISC II 1999), compared with less than 2% in patients with stable CHD (SAPAT 1992). Thus, despite substantial progress in the treatment of ACS with antiplatelet and anti-thrombotic medications (blood thinners), additional therapies are needed to reduce the additional risk associated with unstable CHD. Current guidelines (NCEP 2001) recommend that patients admitted with a major coronary event (MI or ACS) should be considered for treatment with a statin on discharge from the hospital.

Cited advantages of this approach are patient motivation to start therapy at that time and prevention of a "treatment gap" due to inconsistent outpatient follow-up. A previously randomized controlled study of statin therapy in ACS patients (MIRACL study), showed that aggressive cholesterol lowering with atorvastatin 80 mg between 24 and 96 hours after hospital admission in patients with ACS resulted in reduced incidence of recurrent CHD events at 16 weeks. However, the study excluded patients who underwent revascularization (PCI). Thus the study enrolled only a subset of the ACS population.

There is also emerging data from clinical studies supporting the anti-inflammatory actions of statins. One recent randomized controlled study demonstrated that statins decrease the levels of CRP, considered to be a marker of intra-arterial inflammation and a predictor of recurrent adverse cardiovascular events. The relative levels of various lipid measurements, such as LDL-C, triglycerides and HDL-C probably influence the inflammatory and thrombotic (blood clotting) properties, but the exact relationship is not clear. The anti-inflammatory and antithrombotic properties of different statins are likely related to their impact on the lipid profile and their different pleiotropic properties (producing more than one genetic effect).

The present study is designed to compare the effects of rosuvastatin 20 mg versus atorvastatin 80 mg started at maximum 6 days after an ACS to lipid profile (blood cholesterol). Additionally, the hypothesis of beneficial effect on inflammatory markers compared with statins started later will be tested.

c) Summary of study design:

This is a 3-month, randomized, parallel-group study with 2 periods, comparing the efficacy and the safety of rosuvastatin 20 mg versus atorvastatin 80 mg in patients with an acute coronary syndrome (ACS).

* The study comprises a 1st double blind, placebo controlled, period that starts at the admission of the patient for an ACS (clinical symptoms less than 24 hours) until hospital discharge (or a maximum timeline of 6 days).
* The 2nd double blind, double dummy, period starts at Day 0 (i.e. from the hospital discharge or at a maximum of 6 days after admission) and will last 3 months. After validation of eligibility criteria (including a 1st local assessment of CK, creatinine, ALT and an ECG) and the planning of a PCI between 24 hours and 4 days after admission, patients will be randomized into 3 groups:

  1. early started rosuvastatin 20 mg from admission until the end of the study (group 1 - early rosuvastatin 20 mg),
  2. placebo from admission until Day O (i.e. until hospital discharge or for a maximum of 6 days) followed by rosuvastatin 20 mg until the end of the study (group 2 - late rosuvastatin 20 mg),
  3. placebo from admission until Day O (i.e. until hospital discharge or for a maximum of 6 days) followed by atorvastatin 80 mg until the end of the study (group 3 - atorvastatin 80 mg).

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are between 18 and 75 years old
* Patients diagnosed with non ST elevation - acute coronary syndrome (NSTE-ACS)
* Patients with onset of clinical symptoms less than 24 hours prior to their admission for which a PCI is planned or anticipated.

Exclusion Criteria:

* Patients with STEMI (ST elevation myocardial infarction-heart attack) and primary PCI planned within 24 hours of admission will not be included.
* Patients will not be allowed to have taken any cholesterol-lowering medications during 1 month prior to enrolment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of rosuvastatin 20 mg versus atorvastatin 80 mg in measuring ApoB/ApoA ratio at 3 months in acute coronary syndrome patients receiving the study treatment after percutaneous coronary intervention (PCI). | 12 weeks

SECONDARY OUTCOMES:
Efficacy of rosuvastatin 20 mg versus atorvastatin 80 mg in reducing LDL-C 1 month and 3 months post PCI. | 12 weeks
Efficacy of early-started rosuvastatin 20 mg versus placebo on hs-CRP from admission to start of study treatment post PCI. | 12 weeks
Efficacy of rosuvastatin 20 mg versus atorvastatin 80 mg in reducing ApoB/ApoA-1 ratio at 1 month. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A LaHaye, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Vascular Disease Prevention and Research Centre, Hotel Dieu Hospital, Kingston, Ontario